CLINICAL TRIAL: NCT00687934
Title: A Phase 1 Study of the HSP90 Inhibitor, STA-9090, Administered Once-Weekly in Patients With Solid Tumors
Brief Title: Study of STA-9090, Administered Once-Weekly in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-02; 9090-02
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumors
Keywords: metastatic cancer; solid tumor; histologically or cytologically confirmed non-hematological; malignancy that is metastatic or unresectable for which no; standard therapy exists; STA-9090; ganetespib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ganetespib (Experimental): Ganetespib once weekly infusion, dose escalation study, with treatment until progression
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090 — This is a dose-escalation study. The first cohort will consist of three patients who will receive STA 9090 (ganetespib)during a 1-hour infusion once per week for three consecutive weeks followed by a 1 week dose-free interval. Subsequent cohorts will receive higher amounts of STA-9090 (gantespib) provided that the previous dose was well tolerated during cycle 1 (week 1 - 4). Dose escalation will continue until the maximum tolerated dose (MTD) is determined.

SUMMARY:
An open-label dose escalation study of patients with solid tumors treated with STA-9090 (ganetespib)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be documented to be refractory or not candidates for current approved therapies.
* Must have an ECOG status 0-2.
* Peripheral neuropathy < or = 2.
* Must have acceptable organ and marrow function per protocol parameters.
* No clinically significant ventricular arrythmias or ischemia.

Exclusion Criteria:

* Must not be pregnant or breastfeeding.
* Chemotherapy or radiation within 3 weeks.
* Previous radiation to >25% of total bone marrow.
* Previous high dose chemotherapy with autologous or allogeneic hematopoietic stem cell transplantation.
* Primary brain tumors or active brain metastases.
* Use of any investigational agents within 4 weeks.
* Treatment with chronic immunosuppressants.
* Uncontrolled, intercurrent illness.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of STA-9090 (ganetespib) in cancer patients via assessment of dose limiting toxicities | Cycle 1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Premiere Oncology, Santa Monica, California
  - US Oncology Dayton Oncology and Hematology, P.A, Kettering, Ohio

REFERENCES:
- [Derived] Goldman JW, Raju RN, Gordon GA, El-Hariry I, Teofilivici F, Vukovic VM, Bradley R, Karol MD, Chen Y, Guo W, Inoue T, Rosen LS. A first in human, safety, pharmacokinetics, and clinical activity phase I study of once weekly administration of the Hsp90 inhibitor ganetespib (STA-9090) in patients with solid malignancies. BMC Cancer. 2013 Mar 25;13:152. doi: 10.1186/1471-2407-13-152. PMID 23530663